CLINICAL TRIAL: NCT01484769
Title: Method Development and Assessment of the Effects of Tobacco Products on Oral Cavity Cells
Acronym: H&N
Status: Withdrawn | Type: Observational
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Other Study IDs: 360.05
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tissue samples from patients undergoing elective neck dissection will be collected. Primary tumors and adjacent normal tissue from unaffected areas will be collected at the time of surgery. All tissue dissection and removal are part of the standard of care for this type of surgical procedure. Remaining resected tissue will be used for research.
Oversight: Data Monitoring Committee: No

SUMMARY:
Collection of tissues for analysis from patients undergoing elective neck dissection.

The hypothesis of the study is that specific genetic alterations occur in head and neck cancers that have spread to regional and/or distant sites, and these alterations can be identified from biopsy specimens to allow more accurate staging of tumor and better treatment planning.

DETAILED DESCRIPTION:
The standard of care for the treatment of most squamous cell carcinoma of the head and neck is surgical extirpation of the primary tumor and elective neck dissection to remove regional nodes at risk for spread. Via this treatment regimen, the investigators will be able to prospectively obtain tissues for analysis from patients undergoing elective neck dissection.

The specific aims of this study are to compare gene expression between head and neck tumors with and without regional lymph node metastases, and to compare gene expression between head and neck tumor with and without distant metastases.

ELIGIBILITY:
Inclusion Criteria:

* All patients with biochemical evidence of squamous cell carcinoma of the head and neck.

Exclusion Criteria:

* Patients without biomedical evidence of squamous cell carcinoma.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and minors diagnosed with squamous cell carcinoma of the head and neck that will undergo elective neck dissection surgery at either Norton Hospital, Kosair Children's Hospital, or University of Louisville Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-07; Primary Completion 2011-06 (Estimated); Study Completion 2012-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Kosair Children's Hospital, Louisville, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky